CLINICAL TRIAL: NCT00151736
Title: A Randomized, Multi-Center, Phase II Study to Investigate the Safety and Efficacy of SDX-101 (R-etodolac) in Combination With Chlorambucil, and That of Chlorambucil Alone, in Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Safety and Efficacy of SDX-101 (R-Etodolac) in Combination With Chlorambucil, and That of Chlorambucil Alone, in Patients With Chronic Lymphocytic Leukemia (CLL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDX-101-03
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Chlorambucil

ARMS (2):
- Chlorambucil (Experimental): Regime A
  Interventions: Drug: Chlorambucil
- R-etodolac with chlorambucil (Experimental): Regime B
  Interventions: Drug: R-etodolac + chlorambucil

INTERVENTIONS:
Drug: Chlorambucil — Chlorambucil 2mg tablets
  Other Names: SDX-101
  Arms: Chlorambucil
Drug: R-etodolac + chlorambucil — R-etodolac 600mg tablets + chlorambucil 2mg tablets
  Arms: R-etodolac with chlorambucil

SUMMARY:
This is a Phase 2, multi-center, open label, randomized clinical study to evaluate the safety and efficiency of SDX-101 in combination with chlorambucil (CLB) and chlorambucil alone in Chronic Lymphocytic Leukaemia (CLL) patients. The study treatment period will be approximately 24-26 weeks with a follow-up period of approximately 8 weeks. Following the end of treatment, patients with a confirmed complete response, partial response or stable disease will be followed for up to 2 years to assess time to disease progression. Approximately 80 patients with documented diagnosis of B-cell CLL by standard clinical and immunophenotyping criteria will be enrolled into the SDX-101-03 study. This study is being conducted in the following European countries: France, Germany, Poland, Sweden and the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of B-cell CLL by standard clinical and immunophenotypic criteria as specified by the NCI working group revised guidelines for diagnosis and treatment of CLL(32).
2. Binet stages A-C with evidence of active disease requiring treatment by the presence of one or more of the following at the time of study entry:

   * Disease related B symptoms (Fever > 38C [100.5F] for ≥ 2 weeks without evidence of infection, night sweats without evidence of infection, weight loss > 10% within previous 6 mo.).
   * Evidence of progressive marrow failure as manifested by:
   * A decrease in hemoglobin to < 10g/dL, or
   * A decrease in platelet count to < 100 x 10(9)/L within the previous 6 months, or
   * A decrease in absolute neutrophil count (ANC) to < 1.0 x 10(9)/L within 6 months
   * Progressive lymphocytosis with an increase of > 50% over a 2 month period, or an anticipated doubling time of < 6 months.
   * Massive nodes or clusters(i.e., > 10 cm in longest diameter) or progressive lymphadenopathy.
   * Progressive splenomegaly to > 2cm below the left costal margin or other organomegaly with progressive increase over 2 consecutive clinical visits ≥ 2 weeks apart.
3. No prior chemotherapy for CLL.
4. Age ≥ 18 at signing of informed consent.
5. World Health Organization (WHO) performance status ≤ 0-2 (Appendix B).
6. Platelet count > 50,000/μL, hemoglobin > 8.0 g/dl and absolute neutrophil count > 1000/μL.
7. Renal function ≤ 1.5 x upper limit normal (blood urea nitrogen [BUN], serum creatinine)
8. Liver function ≤ 1.5 times upper limit of normal (total bilirubin, SGOT (AST) and SGPT (ALT) values).
9. Female patients of childbearing potential must have a negative pregnancy test (serum or urine Beta-human chorionic gonadotropin, Beta-HCG); men and women of reproductive potential must employ effective contraceptive methods while on study therapy, and for 2 months following completion of treatment.
10. Signed EC/IRB-approved informed consent by patient prior to all study related procedures.

Exclusion Criteria:

1. Active autoimmune manifestation of CLL such as ongoing hemolytic anemia or ITP
2. History of a second malignancy with the exception of cervical cancer,or resected basal cell carcinoma or other malignancies with no evidence of recurrence 5 or more years since diagnosis.
3. Chronic viral infection: positive hepatitis B or hepatitis C serology, known positive for human immunodeficiency virus (HIV) or human T-leukemia/lymphoma virus (HTLV).
4. Transformation to an aggressive B-cell malignancy such as Richter's transformation, prolymphocytic leukemia (PLL) or large B-cell lymphoma.
5. Clinical evidence of CNS involvement with CLL.
6. Serious infection, medical condition, or psychiatric condition that, in the opinion of the investigator, might interfere with the achievement of the study objectives.
7. Treatment with any investigational agent within 4 weeks of study entry.
8. The use of steroids, nonsteroidal anti-inflammatory drugs, regardless of indication (excluding prophylactic use of aspirin for prevention of acute myocardial infarction or stroke)
9. Pregnancy or currently breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2004-09; Primary Completion 2006-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Bone Marrow Biopsy or Aspiration | Baseline + 6 months
  Overall response rate assessment according to National Cancer Institute-Working Group (NCI-WG) criteria using cytogenetic and biomarker evaluations.

SECONDARY OUTCOMES:
Cytogenetic and biomarker evaluations + adverse events | 6 months
  Cytogenetic and biomarker evaluations performed on day 14 (for regimen B) and day 1 (for regimen A) to assess Safety and Tolerability. Study visits to assess safety occur every 2 weeks for 3 months, then every month thereafter. Safety assessments include: medical history, physical examinations, vital sign measurements, adverse event assessment, routine hematology and serum chemistry tests, urinalysis, and ECGs.

CONTACTS AND LOCATIONS:
Locations (22):
- France (2):
  - Chef du Service d'Hematologie Clinique CHU Clemenceau, Caen
  - Service maladies du sang CHRU- rue Michel Polonovski, Lille
- Germany (3):
  - Charité - Benjamin Franklin Medizinische Klinik III Hämatologie, Onkologie und Transfusionsmedizin, Berlin
  - Internistische Schwerpunktpraxis, Erlangen
  - Medizinische Poliklinik der Universität Hämatologie/Onkologie, Würzburg
- Poland (7):
  - Samodzielny Publiczny Szpital Kliniczny AM Klinika Hematologii, Bialystok
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 Akademickie Centrum Kliniczne Akdemii Medycznej w Gdansku Klinika Hematologii, Gdansk
  - Uniwersytet Jagiellonski Collegium Medicum Katedra i Klinika Hematologii, Krakow
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Klinika Hematologii Instytutu Medycyny Wewnetrznej Uniwersytetu Medycznego w Lodzi, Lodz
  - Prywatna Praktyka Lekarska z Osrodkiem Badan Klinicznych Prof. L. Szczepanskiego, Lublin
  - Samodzielny Publiczny Centralny Szpital Kliniczny Katedra i Klinika Hematologii Onkologii i Chorob Wewnetrznych AM, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 Klinika Hematologii, Nowotworow Krwi i Transplantacji Szpiku, Wroclaw
- Sweden (4):
  - Centrum för Hematologi Karolinska Universitetssjukhuset, Solna, Stockholm
  - Hematologkliniken Karolinska Universitetssjukhuset, Huddinge, Stockholm
  - Hematologkliniken Norrlands Universitetssjukhus, Umeå
  - Hematologisektionen Medicincentrum Akademiska sjukhuset, Uppsala
- United Kingdom (6):
  - Royal Bournemouth Hospital Dept. of Haematology, Bournemouth
  - Cardiff and Vale NHS Trust University Hospital of Wales, Cardiff
  - Stobhill Hospital Department of Haematology, Glasgow
  - Leeds General Infirmary Department of Haematology, Leeds
  - Leicester Royal Infirmary Department of Oncology & Haematology, Leicester
  - Nottingham City Hospital NHS Trust, Nottingham